CLINICAL TRIAL: NCT00804284
Title: Post-Licensure Safety Surveillance Study of Routine Use of PENTACEL® Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus b Conjugate (Tetanus Toxoid Conjugate) Vaccine
Brief Title: Database Surveillance Safety Study of PENTACEL® Vaccine
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: M5A11
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Diphtheria; Tetanus; Pertussis; Haemophilus Influenzae
Keywords: DAPTACEL®; PENTACEL®; Diphtheria; Tetanus; Pertussis; Haemophilus influenzae type b
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Haemophilus Infections | interventions — diphtheria-tetanus-five component acellular pertussis-inactivated poliomyelitis -Haemophilus influenzae type b conjugate vaccine; pentacel; Diphtheria-Tetanus-acellular Pertussis Vaccines; PEDIARIX

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pentacel Group: Infants initiated on PENTACEL® vaccine
  Interventions: Biological: DTaP-IPV/Hib
- Other DTap vaccines Group: Infants initiated on other DTaP vaccines
  Interventions: Biological: Other DTap Vaccines

INTERVENTIONS:
Biological: DTaP-IPV/Hib — 0.5 mL, Intramuscular
  Other Names: PENTACEL®
  Groups: Pentacel Group
Biological: Other DTap Vaccines — 0.5 mL, Intramuscular
  Other Names: DAPTACEL®; INFANRIX®; PEDIARIX®; TRIPEDIA®
  Groups: Other DTap vaccines Group

SUMMARY:
The objective for this study is to characterize the safety profile of PENTACEL® vaccine for identification of potential vaccine-related adverse events not currently associated with PENTACEL® vaccine administration.

DETAILED DESCRIPTION:
The study will be conducted at Kaiser Permanente Northern California and will commence with first use of licensed PENTACEL® vaccine within that organization.

Vaccination databases will be reviewed to identify Diphtheria and tetanus toxoid with acellular pertussis (DTaP) vaccinations of accrued subjects. Medical encounter, emergency room, hospitalization, laboratory, state death reporting, and related databases will be reviewed to identify medical care events.

ELIGIBILITY:
Inclusion Criteria:

* Receipt of DTaP vaccine during the study period by a previously unvaccinated child

Exclusion Criteria:

* None

Ages: 6 Weeks to 24 Months | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Receipt of DTaP vaccine during the study period by a previously unvaccinated subjects
Sampling Method: Non-Probability Sample
Enrollment: 62538 (Actual)
Dates: Start 2008-09; Primary Completion 2014-08 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
A summary of all non-elective hospitalization and emergency room visits as well as outcome of interest from chart review. | Up to 6 months post -dose 4 DTap Vaccination
  Outcome of interest identified from Kaiser Permanente Medical Care Program (KPMCP) computerized records via International Classification of Diseases, 9th edition (ICD-9) codes, defined as:
  * Death,
  * Outpatient clinic visit for:
    * seizure occurring within 72 hours of vaccination, Guillain-Barré Syndrome, encephalopathy, encephalitis, alteration of consciousness (other than secondary to another diagnosis), or meningitis
    * hypersensitivity reactions (e.g. urticaria, angioedema, or anaphylaxis) occurring within 72 hours of vaccination,
    * new-onset autoimmune disease (including idiopathic thrombocytopenic purpura, hemolytic anemia).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc
Locations (1):
- Oakland, California, United States

REFERENCES:
- [Derived] Hansen J, Timbol J, Lewis N, Pool V, Decker MD, Greenberg DP, Klein NP. Safety of DTaP-IPV/Hib vaccine administered routinely to infants and toddlers. Vaccine. 2016 Jul 29;34(35):4172-4179. doi: 10.1016/j.vaccine.2016.06.062. Epub 2016 Jun 30. PMID 27373595
- See also: Related Info — http://www.sanofipasteur.com